CLINICAL TRIAL: NCT06880445
Title: Different Perineal Cleaning and Disinfection Preparations Before Vaginal Birth to Maternal/Neonatal Infections and Cost Effectiveness: A Randomized Control Trial
Brief Title: Different Perineal Preparations Before Vaginal Birth to Maternal/Neonatal Infections and Cost Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu-Ying Huang (Other)
Responsible Party: Sponsor-Investigator, Tzu-Ying Huang, Far Eastern Memorial Hospital Deputy Director of Nursing, Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 113236-F
Record Dates: First submitted 2024-12-05; First posted 2025-03-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Perineal Infection; Maternal Infections Affecting Fetus or Newborn; Cost Effectiveness
Keywords: Perineal cleaning and disinfection; Maternal/Neonatal Infections; Cost Effectiveness
MeSH Terms: interventions — Povidone-Iodine; Water

STUDY DESIGN:
Intervention Model Description: This stu dy used the Random Allocation Software developed by Mahmood Saghaei to randomly assign the research subjects into the control group and the experimental group. The control group used clean water to prepare the perineum for the second stage of labor, while the experimental group used betadine disinfection for perineal preparation for the second stage of labor.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perineal Disinfection (Experimental)
  Interventions: Procedure: Povidone-Iodine (PVP-I)
- Perineal Cleaning (Placebo Comparator)
  Interventions: Procedure: Water

INTERVENTIONS:
Procedure: Povidone-Iodine (PVP-I) — The experimental group will use povidone-iodine for disinfection.
  Arms: Perineal Disinfection
Procedure: Water — The control group will undergo perineal preparation using clean water
  Arms: Perineal Cleaning

SUMMARY:
The vaginal microbiome plays a crucial role in women's health, primarily composed of beneficial bacteria such as Lactobacillus, which help maintain an acidic environment in the vagina, preventing the growth of pathogens. Research indicates that the vaginal environment during pregnancy is more conducive to the growth of Lactobacillus. Traditionally, perineal disinfection is performed during vaginal delivery; however, studies have shown that excessive use of disinfectants like povidone-iodine may reduce the presence of Lactobacillus in the vagina. Furthermore, not using perineal disinfection does not increase the risk of postpartum infections for mothers and infants, and may even benefit the development of the newborn's microbiome. Considering the medical costs and nursing labor involved, this study aims to compare the effects of different perineal preparation methods on postpartum infection rates and medical costs, with the goal of improving maternal and infant care quality during delivery and reducing healthcare costs.

5、 Method This study employs an experimental research design. After obtaining informed consent from participants, they will be randomly assigned to either the control group or the experimental group using a random number table. The control group will undergo perineal preparation using clean water, while the experimental group will use povidone-iodine for disinfection. The study will document patient demographics, prenatal vital signs, maternal and infant postpartum temperatures, blood test results, and oral bacterial culture outcomes to monitor postpartum infection rates. The REEDA scale will be used to assess perineal wound healing.

6、Expected results： The anticipated results indicate that using clean water for perineal preparation will not increase the risk of postpartum infections for mothers and infants, while also saving medical costs. Additionally, water disinfection may allow newborns to acquire beneficial bacteria such as Lactobacillus from the mother's vagina during delivery, promoting healthy gut microbiome development.

ELIGIBILITY:
Inclusion Criteria:

Maternity:

* Born after 37 weeks of pregnancy;
* Pregnant women with low-risk pregnancy;
* Be able to communicate in Mandarin and Taiwanese, and be able to read Chinese;
* A single fetus with a cephalic position;
* Aged 18 years or above (inclusive) with clear consciousness and no cognitive impairment;
* Do not use antibiotics during pregnancy;
* There are no fetal diagnostic abnormalities during pregnancy check-up.

Newborn:

* Newborns over 37 weeks
* Apgar Score is greater than 7 points in the first minute of life
* Having given birth to a newborn and undergoing perineal cleaning/disinfection methods specified in the study during the second stage of labor

Exclusion Criteria:

* The mother's water broke for more than 18 hours during labor;
* Mother had a fever;
* Used vacuum suction during delivery;
* Shoulder dystocia;
* Fetal distress;
* A perineal wound of 3 degrees or above

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Different Perineal cleaning and disinfection Preparations Before Vaginal Birth to Maternal/Neonatal Infections and Cost Effectiveness: A Randomized Control Trial | 2Years
  Cases that agree to participate in the study will collect data on a self made login form.
  During the study period, perineal preparation and 24hours postpartum perineal wound healing was assessed using the REEDA scale at the time of discharge and on the day of discharge, and neonatal oral bacterial culture was performed by the researcher.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Banqiao District, Taiwan

IPD SHARING:
Plan to Share IPD: No